CLINICAL TRIAL: NCT02529878
Title: A Prospective Feasibility Study for Convernsion Therapy Using S1/Paclitaxel Chemotherapy Plus Apatinib in Unresectable Gastric Cancer
Brief Title: Study of Convernsion Therapy Using S1/Paclitaxel Chemotherapy Plus Apatinib in Unresectable Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECGC-0001
Record Dates: First submitted 2015-08-19; First posted 2015-08-20 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-02

CONDITIONS: Gastric Cancer
Keywords: gastric caner; Apatinib; S1; conversion therapy; metastatic gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- conversion treatment (Experimental): after 3 cycles S1/Paclitaxel chemotherapy plus Apatinib,subsequent surgery will be conducted with curative intent
  Interventions: Drug: S1/Paclitaxel chemotherapy plus Apatinib

INTERVENTIONS:
Drug: S1/Paclitaxel chemotherapy plus Apatinib — S1:60mg twice daily(after the breakfast and supper) for two weeks, and then suspend for one week Paclitaxel:150mg/m2,iv, 3h, at day1 Apatinib:500mg once daily
  Other Names: SPA

SUMMARY:
The prognosis of metastatic gastric cancer is poor. Chemotherapy occasionally converts an initially unresectable gastric cancer to a resectable cancer. Previous studies showed patients with unresectable gastric cancer may obtain a survival benefit from chemotherapy and subsequent curative surgery. The key of conversion therapy of initially unresectable metastatic GC is the high response rate. Apatinib, a novel targeted inhibitor of VEGF receptor 2 (VEGFR2), shows significant antitumor activity in the patients with GC. The purpose of this study is to investigate the efficacy and safety of S1/Paclitaxel chemotherapy plus Apatinib in the conversion therapys of metastatic gastric cancer.

DETAILED DESCRIPTION:
The investigators will apply SPA regimen for coversional therapy to abtain high response rate.

Paclitaxel：150 mg/m2 i.v.3h , given on the first day. Apatinib, oral ,initial dose :500mg, QD, after meal ( try to take the medicine at the same time of the day ).

Dose adjustment: Down-regulate the dosage to 250 mg per day at the first time. If the patient totally recovers from the toxic reaction after the regulation, we could up-regulate the dosage back to the former level. If the down-regulation occurs again according to the protocol , then the up-regulation will be forbidden.

S-1 dosage: According to the body surface area, the initial dosage of S-1 is decided by the following criteria. Take the medicine twice daily (after breakfast and supper) for 2 weeks, then suspend for 1 week.

Preventive medication: To prevent serious allergic reaction of Paclitaxel, preventive medication should be given in advance. We usually give dexamethasone 20mg orally 12 and 6 hours before the Paclitaxel, and diphenhydramine (or something analogous) 50 mg, cimetidine 300mg (or ranitidine 50mg) I.V. 30-60 minutes before the Paclitaxel.

Repeat the therapeutic schedule every 3 weeks. 3 cycles of neoadjuvant chemotherapy before surgery, stop Apatinib in the last cycle.

3 cycles of adjuvant chemotherapy including S-1 and Apatinib 4 to 6 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* unresectable gastric cancer as proven histologically(AJCC, version 7) under any following condition: unable radical excision due to the local metastasis of invasion metastasis to the lymph node beside the abdominal aorta, non-extensive metastasis to liver( not more than three metastatic foci of radical excision), Peritoneal metastasis(CY1,P1,P2), kukerburg tumor
* Definitely diagnosed as above stage of gastric cancer before operation via CT of MRI, ultrasonic endoscopy, PET-CT, or through the laparoscopic exploration if necessary
* Untreated(e.g. radiotherapy, chemotherapy, target therapy and immunotherapy)
* Negative HER-2 state
* ECOG(Eastern Cooperative Oncology Group) :0~2
* Age: 18~75 years old
* Normal hemodynamic indices before the recruitment(including blood cell count and liver/kidney function ). For example: WBC>4.0*109/L, NE>1.5*109/L, PLT>100*109/L, BIL<1.5 times of upper limit of normal reference value, ALT and AST<2.5 times of upper limit of normal reference value, and CRE<1.2mg/dl
* Good cardiac function before the recruitment, no seizure of myocardial infarction in past half years, and controllable hypertension and other coronary heart disease
* Not concomitant with other uncontrollable benign disease before the recruitment(e.g. the infection in the kidney, lung and liver)
* Not participating in other clinical trials before and during the treatment
* Signed the Informed Consent Form

Exclusion Criteria:

* not conforming above inclusion conditions
* Distal metastasis to lung, brain, and bone
* Ever operation on the stomach
* Operation intolerance due to other systemic basic disease
* Ever administrated with other drugs(including TCM drugs) before the recruitment, or no guarantee of progress according to the study requirement after recruitment
* Allergy to the drugs in this protocol
* Pregnant and lactating women
* Women at childbearing age and of pregnancy desire during the study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
radical resection rate | 4 months
  the radical resection rates

SECONDARY OUTCOMES:
overall survival | 3 years
  the overall survival time
adverse events | 6 months
  number and degree of adverse events
reaction rate | 4 months
  the reaction rate of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Xiangdong Cheng, MD, Principal Investigator — The First Affiliated Hospital of Zhejiang Chinese Medical University
Locations (1):
- the First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China